CLINICAL TRIAL: NCT01017861
Title: The Effect of Pregnancy on Temporal Summation and Venipuncture Pain Perception
Status: Completed | Type: Observational
Sponsor: Samuel Lunenfeld Research Institute, Mount Sinai Hospital (Other)
Responsible Party: Dr. Jose Carvalho, Mount Sinai Hospital
Other Study IDs: 09-04
Record Dates: First submitted 2009-11-19; First posted 2009-11-23 (Estimated); Last update posted 2010-09-28 (Estimated); Status verified 2010-09

CONDITIONS: Pain; Pregnancy
Keywords: Temporal summation; Venipuncture pain
MeSH Terms: conditions — Pain

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (4):
- Pregnant, 12th week: Pregnant women in the 12th week of pregnancy.
- Pregnant, 28th week: Pregnant women in the 28th week of pregnancy.
- Pregnant, full term: Pregnant women at full term, in hospital for an elective cesarean section.
- Non pregnant women: Non pregnant women

SUMMARY:
Recent studies have shown that women are more likely to experience pain in many medical situations. During pregnancy, women may experience an increase in pain threshold. This is thought to be related to hormonal changes and an increase in the level of certain natural pain-relieving substances in their bodies.

It is important to develop simple tests to identify woman at higher risk for pain so the investigators can help them.

Temporal summation is what happens when a person becomes more sensitive to a certain feeling on their skin when it is applied several times over the course of several seconds. The investigators hypothesize that pregnant women show decreased temporal summation and pain scores to venipuncture, compared to non-pregnant women.

DETAILED DESCRIPTION:
Recent epidemiologic studies have shown that women are at substantially greater risk for many clinical pain conditions, and there is a suggestion that postoperative and procedural pain may be more severe among women then men. During pregnancy, women experience an elevation in the threshold to pain and discomfort. In addition to hormonal changes, the changes in pain perception during pregnancy may be related to an increase in endogenous opioids.

Pain is the most feared experience in the intra and postpartum period, and severe pain experienced during this time can lead to significant morbidity, including chronic pain and depression. Much attention has been paid to tests that can predict patients at higher risk for pain. Temporal summation (TS) has been shown to be a simple and reliable test. Temporal summation represents the physiological wind-up phenomenon taking place at the spinal level of the central pain pathways. TS extent can be measured in humans by administering a series of noxious stimuli of constant intensity and of various modalities in order to evoke an increase in perceived pain. It is a very simple and easy test to perform, and very well tolerated by patients. Whether TS changes in pregnancy and whether TS in pregnancy correlates with pain perception during acute stimuli such as venipuncture is unknown.

ELIGIBILITY:
Inclusion Criteria:

* informed consent
* able to communicate in English
* healthy pregnant patients in the 1st, 2nd and 3rd trimesters
* healthy non-pregnant patients

Exclusion Criteria:

* refusal to participate
* Patients under age 18 or over age 40
* Inability to communicate in English
* Use of analgesics, anti-depressants and muscle relaxants
* self-report of substance abuse
* previous injury to the non-dominant arm/forearm

Ages: 18 Years to 40 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Pregnant patients presenting at the venipuncture clinic for routine bloodwork throughout their pregnancy.
  Full term pregnant patients admitted to the hospital for and elective cesarean section.
  Non pregnant volunteers.
Sampling Method: Probability Sample
Enrollment: 80 (Estimated)
Dates: Start 2009-10; Primary Completion 2010-01 (Actual); Study Completion 2010-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jose Carvalho, MD, Principal Investigator — MOUNT SINAI HOSPITAL
Locations (1):
- Mount Sinai Hospital, Toronto, Ontario, Canada